CLINICAL TRIAL: NCT06414772
Title: Evaluation of an Electronic Tool Designed to Facilitate Communication Between Allophone Patients or Patients With Communication Difficulties and Physicians in Pediatric Emergency Departments.
Brief Title: Evaluation of an E-tool Designed to Facilitate Communication Between Allophone Patients and Pediatricians in Emergency Departments.
Acronym: ENTENTE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022/739
Record Dates: First submitted 2024-01-10; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Language Barrier
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With MARTI e-tool (Experimental)
  Interventions: Other: Use of MARTI application in addition with a classical consultation/support
- Without MARTI e-tool (No Intervention)

INTERVENTIONS:
Other: Use of MARTI application in addition with a classical consultation/support — Participants will use MARTI in order to establish the medical history during their waiting time.
  Arms: With MARTI e-tool

SUMMARY:
In France, over 21 million people visit emergency departments every year, 10% of whom speak little or no French. The language barrier is a problem for patient safety and quality of care. Ethical and financial aspects are also affected. Unnecessary tests are more frequent, hospital stays more numerous and longer. Patient's management may be inappropriate. Patients are less satisfied, understand and adhere less to cmanagement and recommendations.

Some solutions are available to the emergency physician, but their contribution is limited. A professional interpreter is reliable and takes cultural aspects into account, but his or her cost is high and availability incompatible with emergency care. Translation by a close relative poses the problem of confidentiality. Telephone interpreting is available at any time, but is expensive and less satisfying than direct interaction. Computerized machine translation is economical and easy to access, but does not take into account all medical terms. It also poses a data protection problem. Phraselators translate predefined phrases with precision, but are time-consuming and unsophisticated.

In addition, these aids are used during the consultation. They are therefore difficult to combine and take up care time.

This care time is mainly devoted to establishing medical history essential for the diagnosis, prognosis and treatment decisions.

MARTI is a digital tool for pediatric emergency room consultations. Its aim is to enable the emergency physician to start the consultation with a medical history completed autonomously by the parents during their waiting time. Its content has been developed by emergency physicians.

Language and cultural barriers are overcome through the use of simple phrases and pictograms developed with linguists, language schools and Immigrant organizations.

MARTI was used in a pediatric emergency department. Feedback from patients and carers indicates that it is ready to be tested in real-life conditions.

This pilot study is designed to evaluate how MARTI improves communication with an allophone or a person with comprehension difficulties, according to the emergency physician in charge of the consultation.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Person responsible for a child admitted to pediatric emergency.
* Person with a language barrier.
* Person speaking one of the 11 languages proposed by MARTI.
* Signed informed consent indicating that the subject has understood the purpose and procedures of the study and agrees to participate in the study and to abide by the requirements and restrictions inherent in the study.
* Affiliation with a health insurance

Exclusion Criteria:

* Person who shares a common language with the physician.
* Illiterate person.
* Person accompanying a child with a life-threatening emergency.
* Subject without health insurance.
* Pregnant women.
* Subject in the exclusion period of another study or in the "national volunteer file".

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Quality of communication | Day 1
  The quality of communication will be assessed using a Likert-type scale to be completed by the emergency physician at the end of the consultation (whether MARTI was used or not).
  Originally, Likert scale is a rating scale that assesses opinions, attitudes, or behaviors quantitatively in five point expressed as follows: strongly agree, agree, neutral, disagree, strongly disagree. These points have been kept for the scale of the study, which was adapted with items like "Using MARTI app reduced my anxiety" (for caregivers), "The app is easy to use" (for parents), etc.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Besançon, Besançon
  - Hôpital Nord Franche-Comté, Trévenans

IPD SHARING:
Plan to Share IPD: No